CLINICAL TRIAL: NCT02935283
Title: Neuroimaging and Neuropsychological Outcomes in Urea Cycle Disorders
Acronym: UCD
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Andrea Gropman, Chief, Division of Neurogenetics and Developmental Pediatrics, Children's National Research Institute
Other Study IDs: UCD 5113
Record Dates: First submitted 2016-05-12; First posted 2016-10-17 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- OTCD participants: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD who can undergo MRI and behavioral testing
  Interventions: Procedure: MRI; Behavioral: Behavioral
- Normal controls: Healthy males or females without known medical or metabolic disorder (control group) who can undergo MRI and behavioral testing
  Interventions: Procedure: MRI; Behavioral: Behavioral
- HA recovery group: Female carriers of ornithine transcarbamylase deficiency (OTCD) or males with late onset presentation of OTCD or participants with CPS-1 who have had a recent hyperammonemic episode who can undergo MRI and behavioral testing
  Interventions: Procedure: MRI; Behavioral: Behavioral
- Distal UCD: Males and females with ASSD and ASLD who can undergo MRI and behavioral testing
  Interventions: Procedure: MRI; Behavioral: Behavioral

INTERVENTIONS:
Procedure: MRI — MRI, fMRI, 1H MRS, DTI
Behavioral: Behavioral — Battery of executive function tasks
  Other Names: cognitive testing, Neuropsychological testing

SUMMARY:
In proximal urea cycle disorders (UCD), particularly ornithine transcarbamylase deficiency (OTCD), hyperammonemia (HA) causes increased brain glutamine (Gln) which perturbation is thought to be at the core of the neurological injury. In contrast, in distal UCD such as citrullinemia (argininosuccinate synthetase deficiency; (ASSD) and argininosuccinic aciduria (argininosuccinate lyase deficiency); (ASLD) cognitive impairment and neuropsychiatric disease are common even in the absence of acute HA. As a consequence, both citrulline and argininosuccinate (ASA) or their metabolic products have been implicated as neurotoxic. In this project the investigators will use state-of- the-art neuroimaging and neuropsychological methods to investigate whether patients with OTCD have chronically elevated brain Gln and reduced myo-inositol (mI) levels that correlate with regional brain structural abnormalities and neurocognitive dysfunction. The researchers will further investigate whether during an acute episode of HA elevated brain Gln and decreased mI levels correlate with the magnitude of cytotoxic edema and whether a Gln/mI ratio threshold can be identified at which the cytotoxic edema is followed by cell loss. Finally, the researchers will investigate whether regions of brain damage in ASSD and/or ASLD are distinct from those in OTCD and compare brain Gln levels in ASSD and ASLD in the absence of HA to those in OTCD. The investigators will also seek to determine if brain citrulline and ASA can be identified in the brains of patients with distal UCD and whether they correlate with brain abnormalities seen in MRI and neuropsychological testing. This project will elucidate the chronology of brain pathology both in acute hyperammonemia and chronic UCD and whether, proximal and distal UCD differ in their pathophysiology of brain damage.

DETAILED DESCRIPTION:
UCDs are a group of rare genetic diseases that affect how protein is broken down in the body. The cause of UCDs is a deficiency in one of eight enzymes responsible for removing ammonia, a waste product of protein metabolism, from the bloodstream. Normally, ammonia is converted into urea and then removed from the body in the form of urine. However, in people with UCDs, ammonia accumulates unchecked and is not removed from the body. Toxic levels of ammonia can build up and cause irreversible neurologic damage that can affect metabolism, cognition, sensation, and movement. This study will focus on the most common enzyme disorder among UCDs, ornithine transcarbamylase deficiency (OTCD), a disorder inherited from mothers. Using different types of magnetic resonance imaging (MRI), this study will evaluate how UCD-related neurologic injuries affect metabolism, cognition, sensation, and movement in adults with OTCD.

This study will be separated into three sections. The first study will study longitudinal changes in OTCD. The second section will study the recovery of OTCD participants from a hyperammonemic episode over time. The third section will be a longitudinal study of the distal urea cycle disorders. In all cases, participants in this study will attend an initial study visit that will include a review of medical history, current symptoms, impairments, and diet history; a physical exam; a full neurological exam; and cognitive and motor testing. During this visit, participants will undergo imaging studies and additional cognitive and motor testing over a 1-2-day period. This will include standard MRI studies and four sessions consisting of functional MRI (fMRI) (CNMC only), diffusion tensor imaging, and 1H magnetic resonance spectroscopy. For the fMRI study, participants perform various motor and behavioral tasks while in the imaging scanner. Magnetic resonance spectroscopy (MRS) is used to study and evaluate the chemical makeup of specific brain areas. Diffusion tensor imaging is used to assess myelination of major brain pathways and their alteration in disease states. This study will involve multiple time point participation. The study will be conducted at Children's National Medical Center and Boston Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for group 1:

1. Confirmed diagnosis of ornithine transcarbamylase deficiency (OTCD) by genetic analysis (genotype) and/or enzyme analysis with at least a single episode of HA hyperammonemic (HA) encephalopathy
2. Ability to undergo MRI without sedation
3. Ages 7 - 50 years
4. Ability to provide informed consent or assent to the procedures
5. Healthy controls (age and gender matched)

Inclusion criteria for group 2:

1. Males and females with a UCD who are having an acute metabolic crisis, with ammonia levels between 100-300 µM
2. Subjects must be awake, and not comatose and able to maintain patent airway on their own and in the opinion of the examining physician, medically stable without risk for acute decompensation and must continue to be stable based on visual contact, vital sign measurement and voice contact with subjects while in the scanner
3. Age range 7-30 years
4. Able to undergo neuroimaging safely (i.e. without ferromagnetic devices)
5. Sexually active female of childbearing potential must agree to urine pregnancy test
6. Admitted to the hospital for treatment of HA at one of the 4 sites for this study
7. Can be subjects who were originally enrolled in aim 1 who then have HA (they will cross over to aim 2)

Inclusion criteria for group 3

1. Confirmed diagnosis of arginosuccinate ASSD, and ASLD by genotype and/or enzyme analysis or healthy age and gender matched control
2. Ability to undergo MRI without sedation
3. Age 7 - 30 years
4. Able to provide informed consent or assent to the procedures

Exclusion Criteria:

Exclusion Criteria for group 1:

1. Inability to undergo MRI without sedation
2. Metal implants, including orthodontic braces
3. Other health conditions contra-indicated in MRI
4. Medically unstable at time of scheduled research visit
5. Unable to provide informed consent or assent to the procedures

Exclusion criteria for group 2:

1. Ammonia level > 300 µM, or <100 µM
2. Presence of coma and/or inability to maintain a patent airway
3. Age <7 or >30 years
4. Subject with ferromagnetic device that precludes safe MRI imaging
5. Pregnant female
6. Unstable medically, at risk for decompensations
7. Combative, or severely neurologically compromised irrespective of ammonia level and showing declining medical status in the scanner based on visual, voice contact and electronic HR monitoring.

Subjects must be awake, and not comatose and able to maintain patent airway on their own

Exclusion criteria for group 3:

1. Inability to undergo MRI without sedation
2. Metal implants, including orthodontic braces
3. Other health conditions contra-indicated for MRI
4. Medically unstable at time of scheduled research visit
5. Unable to provide informed consent or assent

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants have a urea cycle disorder or are healthy controls ages 7-30 years, male and female. Participants who have had a recent hyperammonemic episode are eligible for a more detailed analysis.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2016-08; Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Concentration of Glutamine and Myoinositol by MRS | baseline and 2year follow up
  Concentration based on area under curve on 1H MRS and quantitated by LCModel. A metabolite's tissue concentration is related to the integrated amplitude of the MRS signal it produces. Integrated amplitude is the area under the MRS signal curve. While MRS signals are usually acquired in the time domain as free induction decays or echoes, they are usually viewed and analyzed in the frequency domain. The frequency domain representation is derived from the acquired time domain data by the Fourier Transform. The protocols used selects 257 averages. This means, 257 free induction decays. The machine summates the data at each time point to generate one value for the area under the curve. Therefore, we don't have the measurement at each time point.
  Furthermore, we measured voxels in two different brain areas containing different kinds of brain matter: one voxel was located in posterior cingulate gray matter (PCGM) and the other in parietal white matter (PWM).
Change in Fractional Anisotropy | baseline and 2 year follow up
  Measure of white matter integrity in OTCD Patients and Controls in frontal white matter. Fractional anisotropy values fall on a scale of 0 to 1, with 0 meaning that the diffusion of water is isotropic and unrestricted, or equally restricted, in all directions and with 1 meaning that diffusion occurs along only one axis and is fully restricted along all other directions. Scores closer to 1 are associated with intact white matter while scores closer to 0 are associated with white matter damage.

SECONDARY OUTCOMES:
Change in behavioral testing results | baseline and 2 year follow up
  correlation of the findings from neuroimaging with cognitive functioning that assesses executive function

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Gropman, M.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be kept on UCD website and released after study completion
Supporting Information: Study Protocol, CSR
Time Frame: One year after study completion and available for 5 years

REFERENCES:
- [Result] Pacheco-Colon I, Washington SD, Sprouse C, Helman G, Gropman AL, VanMeter JW. Reduced Functional Connectivity of Default Mode and Set-Maintenance Networks in Ornithine Transcarbamylase Deficiency. PLoS One. 2015 Jun 11;10(6):e0129595. doi: 10.1371/journal.pone.0129595. eCollection 2015. PMID 26067829
- [Result] Sprouse C, King J, Helman G, Pacheco-Colon I, Shattuck K, Breeden A, Seltzer R, VanMeter JW, Gropman AL. Investigating neurological deficits in carriers and affected patients with ornithine transcarbamylase deficiency. Mol Genet Metab. 2014 Sep-Oct;113(1-2):136-41. doi: 10.1016/j.ymgme.2014.05.007. Epub 2014 May 20. PMID 24881970
- [Result] Gropman AL, Shattuck K, Prust MJ, Seltzer RR, Breeden AL, Hailu A, Rigas A, Hussain R, VanMeter J. Altered neural activation in ornithine transcarbamylase deficiency during executive cognition: an fMRI study. Hum Brain Mapp. 2013 Apr;34(4):753-61. doi: 10.1002/hbm.21470. Epub 2011 Nov 23. PMID 22110002
- [Result] Gropman AL, Gertz B, Shattuck K, Kahn IL, Seltzer R, Krivitsky L, Van Meter J. Diffusion tensor imaging detects areas of abnormal white matter microstructure in patients with partial ornithine transcarbamylase deficiency. AJNR Am J Neuroradiol. 2010 Oct;31(9):1719-23. doi: 10.3174/ajnr.A2122. Epub 2010 May 20. PMID 20488904
- [Result] Oldham MS, VanMeter JW, Shattuck KF, Cederbaum SD, Gropman AL. Diffusion tensor imaging in arginase deficiency reveals damage to corticospinal tracts. Pediatr Neurol. 2010 Jan;42(1):49-52. doi: 10.1016/j.pediatrneurol.2009.07.017. PMID 20004862
- [Result] Gropman AL, Fricke ST, Seltzer RR, Hailu A, Adeyemo A, Sawyer A, van Meter J, Gaillard WD, McCarter R, Tuchman M, Batshaw M; Urea Cycle Disorders Consortium. 1H MRS identifies symptomatic and asymptomatic subjects with partial ornithine transcarbamylase deficiency. Mol Genet Metab. 2008 Sep-Oct;95(1-2):21-30. doi: 10.1016/j.ymgme.2008.06.003. Epub 2008 Jul 26. PMID 18662894
- [Result] Shapiro E, Bernstein J, Adams HR, Barbier AJ, Buracchio T, Como P, Delaney KA, Eichler F, Goldsmith JC, Hogan M, Kovacs S, Mink JW, Odenkirchen J, Parisi MA, Skrinar A, Waisbren SE, Mulberg AE. Neurocognitive clinical outcome assessments for inborn errors of metabolism and other rare conditions. Mol Genet Metab. 2016 Jun;118(2):65-9. doi: 10.1016/j.ymgme.2016.04.006. Epub 2016 Apr 14. PMID 27132782
- [Result] Waisbren SE, He J, McCarter R. Assessing Psychological Functioning in Metabolic Disorders: Validation of the Adaptive Behavior Assessment System, Second Edition (ABAS-II), and the Behavior Rating Inventory of Executive Function (BRIEF) for Identification of Individuals at Risk. JIMD Rep. 2015;21:35-43. doi: 10.1007/8904_2014_373. Epub 2015 Feb 25. PMID 25712381
- [Result] Seminara J, Tuchman M, Krivitzky L, Krischer J, Lee HS, Lemons C, Baumgartner M, Cederbaum S, Diaz GA, Feigenbaum A, Gallagher RC, Harding CO, Kerr DS, Lanpher B, Lee B, Lichter-Konecki U, McCandless SE, Merritt JL, Oster-Granite ML, Seashore MR, Stricker T, Summar M, Waisbren S, Yudkoff M, Batshaw ML. Establishing a consortium for the study of rare diseases: The Urea Cycle Disorders Consortium. Mol Genet Metab. 2010;100 Suppl 1(Suppl 1):S97-105. doi: 10.1016/j.ymgme.2010.01.014. Epub 2010 Feb 10. PMID 20188616
- [Result] Jan W, Zimmerman RA, Wang ZJ, Berry GT, Kaplan PB, Kaye EM. MR diffusion imaging and MR spectroscopy of maple syrup urine disease during acute metabolic decompensation. Neuroradiology. 2003 Jun;45(6):393-9. doi: 10.1007/s00234-003-0955-7. Epub 2003 May 8. PMID 12736767